CLINICAL TRIAL: NCT04458363
Title: Convalescent Plasma to Optimize Treatment of COVID-19 Disease in Pediatric Patients: A Feasibility Study
Brief Title: Convalescent Plasma in Pediatric COVID-19
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Preeti Jaggi, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000789
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: COVID
Keywords: COVID-19; Pediatric; Convalescent Plasma; Safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (CP) (Experimental): Once the patient meets criteria for CP infusion (severity of disease and risk factor determination and absence of exclusion criteria) convalescent plasma will be administered
  Interventions: Biological: Convalescent Plasma (CP); Drug: Standard COVID-19 therapies

INTERVENTIONS:
Biological: Convalescent Plasma (CP) — Once the patient meets criteria for CP infusion (severity of disease and risk factor determination and absence of exclusion criteria), an ABO compatible product will be identified. The CP dose administered will be 10mL/kg/dose (up to 2 units per dose) times two doses per patient for a total dose of 20 mL/kg. Patients will be followed for adverse events and clinical response. Research blood testing will be obtained prior to infusion (baseline) and serially weekly afterwards until clinical resolution. Patients will receive 2 doses equaling 20 mL/kg (if available) of ABO compatible CP over 24-48 hours if they do not experience grade 3-5 adverse events that are possible, probably, or definitely attributed to CP after the first dose. Patients will be followed for adverse events for a minimum of 28 days after the last infusion of CP.
Drug: Standard COVID-19 therapies — If clinical status permits, administration of additional COVID-19 therapies should be delayed 48 hours or more from CP infusion completion. Supportive care will be administered by best clinical practice.

SUMMARY:
COVID-19 is increasingly affecting children but convalescent plasma (CP) has not been adequately studied in children to date. The study will determine safety of convalescent plasma for pediatric patients with severe, or at high risk for severe, COVID-19 disease.

DETAILED DESCRIPTION:
COVID19 is an emerging infection with no current approved treatment or prevention. COVID-19 is increasingly affecting children but convalescent plasma (CP) has not been adequately studied in children to date. The study will determine safety of convalescent plasma for pediatric patients with severe, or at high risk for severe, COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0 to 22 years of age
* SARS-CoV-2 infection documented by RNA RT-PCR detection
* Admitted to an acute care facility
* Ability of patient or guardian to provide consent and assent (if applicable); if patient is intubated assent may be waived

Exclusion Criteria:

* Pregnancy/ breast feeding
* Medical condition that increases the risk of plasma infusion
* Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products).

Inclusion criteria for infusion:

* Severe COVID-19 disease, OR
* Moderate disease with a risk of progression to severe or life threatening disease, OR
* Severely immunocompromised patient with any illness attributed to COVID-19 disease requiring inpatient care.

Exclusion to infusion:

* Pregnancy/ breast feeding
* Medical condition that increases the risk of plasma infusion
* Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products).

Ages: 0 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Number of grade 3-5 adverse events that are possible, probably or definitely related to the convalescent plasma (CP) infusion | 28 days
  Safety of convalescent plasma for pediatric patients will be determined by capturing the grade 3-5 adverse events that are possible, probably or definitely related to the CP infusion, defined using the NCI Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Change in percent of supplemental oxygen | Baseline, 72 hours after infusion
  Change in percent of supplemental oxygen within 72 hours after infusion
Number of patients that required change in level of respiratory support | Baseline, 72 hours after infusion
  Number of patients that required change in level of respiratory support such as nasal canula, non-invasive ventilation, mechanical ventilation, high frequency oscillator ventilation, and extracorporeal membrane oxygenation (ECMO)
Mortality | up to 1 year
  Number of deaths
Mean length of ICU stay (days) | Up to 28 days
  Length of ICU stay (days) will be recorded
Mean length of hospital stay (days) | Up to 28 days
  Length of hospital stay (days) will be recorded
Mean length of ventilation (days) | Up to 28 days
  Length of ventilation (days) will be recorded
Number of patients with progression to renal dysfunction and/or multisystem organ failure | up to 1 year
  Number of patients with progression to renal dysfunction and/or multisystem organ failure will be recorded
IL-6 level | up to 28 days
  Cytokine milieu will be assayed by Luminex
Number of anti-SARS CoV 2 specific T cells | up to 28 days
  Cellular studies will be used for evaluation of anti-SARS CoV 2 specific T cells
Diversity of circulating T cells | up to 28 days
  Cellular studies will be used for evaluation of diversity of circulating T cells
ARS-CoV-2 Antibody Titer | up to 28 days
  Antibody titers to SARS-CoV-2 evaluation will be performed in vivo
SARS-CoV-2 Neutralizing Titer | up to 28 days
  Neutralizing antibodies are a type of virus specific antibody that not only bind virus but bind in a manner that prevents viral infection. Test will be will be performed in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Jaggi, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No